CLINICAL TRIAL: NCT03867396
Title: Evaluation of Speech-in-noise Performance in Cochlear Implant Recipients Using Either a Conventional Hearing Aid or a CROS Device on the Contralateral Ear
Brief Title: Evaluation of Speech-in-noise Performance in Cochlear Implant Recipients With a CROS Device on the Contralateral Ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-1101
Record Dates: First submitted 2019-02-19; First posted 2019-03-08 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Cochlear Implant; Hearing Loss; Hearing Aids; Hearing Tests
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss | interventions — Hearing Aids; Cochlear Implants

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into a group where they wear one of the processors and the order of conditions will be assessed, then they will switch to wear the other processor and the order of conditions will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cochlear Implant and Hearing Aid (Active Comparator): Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests.
  Interventions: Device: Hearing Aid
- Cochlear Implant alone (Active Comparator): Subject only uses the cochlear implant; hearing on the contralateral side is unaided.
  Interventions: Other: Cochlear Implant Alone
- Cochlear Implant and CROS (Experimental): Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device.
  Interventions: Device: CROS

INTERVENTIONS:
Device: CROS — Advanced Bionics CROS
  Arms: Cochlear Implant and CROS
Device: Hearing Aid — Advanced Bionics Naida hearing aid
  Arms: Cochlear Implant and Hearing Aid
Other: Cochlear Implant Alone — No hearing device on contralateral ear
  Arms: Cochlear Implant alone

SUMMARY:
Speech understanding in noise remains the greatest challenge for people using cochlear implants, particularly when the speech of interest comes from the side of the head opposite to the implant. Recent findings in hearing technology allow for people to either use a hearing aid or a Contralateral Routing of Signal (CROS) device on the non-implanted ear. Differences in speech understanding may result depending on the device chosen by a person, and these differences may be measureable through speech discrimination measurement methods.

This study intends to determine whether or not a CROS device improves speech perception in noise when the source of the speech of interest originates from the side of the head opposite to the implant.

ELIGIBILITY:
Inclusion Criteria*:

* An Advanced Bionics cochlear implant recipient with at least 6 months of listening experience
* Low frequency Pure Tone Audiometry (PTA)

Exclusion Criteria*:

* Non-English speakers

  * Additional Inclusion and Exclusion criteria apply

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Anderson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with Advanced Bionics.
Supporting Information: Study Protocol, SAP
Time Frame: From first patient through Institutional Review Board (IRB) study close.
Access Criteria: The de-identified data will be shared to with Advanced Bionics in a password protected Excel sheet downloaded from research database.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cochlear Implant (CI) and Hearing Aid, Then CI and CROS, Then CI Alone: 1. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests. Hearing Aid: Advanced Bionics Naida hearing aid.
  2. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
  3. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
- Cochlear Implant (CI) and Hearing Aid, Then CI Alone, Then CI and CROS: 1. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests.Hearing Aid: Advanced Bionics Naida hearing aid.
  2. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
  3. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
- Cochlear Implant (CI) and CROS, Then CI and Hearing Aid, Then CI Alone.: 1. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
  2. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests. Hearing Aid: Advanced Bionics Naida hearing aid.
  3. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
- Cochlear Implant (CI) and CROS, Then CI Alone, Then CI and Hearing Aid: 1. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
  2. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
  3. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests. Hearing Aid: Advanced Bionics Naida hearing aid.
- Cochlear Implant (CI) Alone, Then CI and CROS, Then CI and Hearing Aid: 1. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
  2. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
  3. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests. Hearing Aid: Advanced Bionics Naida hearing aid.
- Cochlear Implant (CI) Alone, Then CI and Hearing Aid, Then CI and CROS: 1. Subject only uses the cochlear implant; hearing on the contralateral side is unaided. Cochlear Implant Alone: No hearing device on contralateral ear.
  2. Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests. Hearing Aid: Advanced Bionics Naida hearing aid.
  3. Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device. CROS: Advanced Bionics CROS.
Period: Intervention 1
Arm/Group | Cochlear Implant (CI) and Hearing Aid, Then CI and CROS, Then CI Alone | Cochlear Implant (CI) and Hearing Aid, Then CI Alone, Then CI and CROS | Cochlear Implant (CI) and CROS, Then CI and Hearing Aid, Then CI Alone. | Cochlear Implant (CI) and CROS, Then CI Alone, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and CROS, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and Hearing Aid, Then CI and CROS
Started | 8 | 8 | 7 | 5 | 7 | 5
Data Collection | 8 | 5 | 7 | 5 | 0 | 0
Completed | 8 | 5 | 7 | 5 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 7 | 5
Period: Intervention 2
Arm/Group | Cochlear Implant (CI) and Hearing Aid, Then CI and CROS, Then CI Alone | Cochlear Implant (CI) and Hearing Aid, Then CI Alone, Then CI and CROS | Cochlear Implant (CI) and CROS, Then CI and Hearing Aid, Then CI Alone. | Cochlear Implant (CI) and CROS, Then CI Alone, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and CROS, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and Hearing Aid, Then CI and CROS
Started | 8 | 5 | 7 | 5 | 0 | 0
Completed | 8 | 5 | 7 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Cochlear Implant (CI) and Hearing Aid, Then CI and CROS, Then CI Alone | Cochlear Implant (CI) and Hearing Aid, Then CI Alone, Then CI and CROS | Cochlear Implant (CI) and CROS, Then CI and Hearing Aid, Then CI Alone. | Cochlear Implant (CI) and CROS, Then CI Alone, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and CROS, Then CI and Hearing Aid | Cochlear Implant (CI) Alone, Then CI and Hearing Aid, Then CI and CROS
Started | 8 | 5 | 7 | 5 | 0 | 0
Completed | 8 | 5 | 7 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographics data and baseline measurements were only collected for participants who completed the study.
Groups:
- All Participants: All participants in crossover study.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Implant Side [Count of Participants; unit: Participants]
  Left | 9
  Right | 16
Implant Device [Count of Participants; unit: Participants]
  HiRes Ultra with HiFocus Mid-Scal | 4
  HiRes Ultra with HiFocus 1J | 8
  HiRes 90K | 12
  CII Bionic Ear | 1
Contralateral Ear Device [Count of Participants; unit: Participants]
  Nothing | 5
  Hearing Aid | 19
  Contralateral Routing of Signal (CROS) device | 1
Has Tinnitus [Count of Participants; unit: Participants]
  Tinnitus | 14
  No Tinnitus | 10
  Unknown | 1
Tinnitus Frequency [Count of Participants; unit: Participants]
  Constant | 7
  Intermittent | 6
  Not Sure | 1
  Missing | 11
Tinnitus Ears [Count of Participants; unit: Participants]
  Right | 2
  Left | 1
  Both | 8
  Not Sure | 3
  None/Missing | 11
Exposure to Excessive Noise [Count of Participants; unit: Participants]
  Exposure to Excessive Noise | 11
  No Exposure to Excessive Noise | 14
Ear Protection with Excessive Noise [Count of Participants; unit: Participants]
  Ear Protection | 3
  No Ear Protection | 8
  Missing | 14
Head Trauma [Count of Participants; unit: Participants]
  Head Trauma | 3
  No Head Trauma | 21
  Missing | 1
Cognition/Memory Concern [Count of Participants; unit: Participants]
  Cognition/Memory Concern | 3
  No Concern | 21
  Missing | 1
Diagnosis Related to Cognition/Memory [Count of Participants; unit: Participants]
  Has Diagnosis Related to Cognition/Memory | 2
  No Diagnosis Related to Cognition/Memory | 22
  Missing | 1
Hearing loss duration (years) [Mean (Standard Deviation); unit: years] — Population: Data was not collected for one participant
  years
    number analyzed (Participants) | 24
    (all) | 29.7 (16.6)
Years since first hearing aid fit [Mean (Standard Deviation); unit: years] — Population: Data was not collected for one participant
  years
    number analyzed (Participants) | 24
    (all) | 20.8 (14.4)
Daily Use of Implant (hours) [Mean (Standard Deviation); unit: hours] — Population: Data was not collected for 4 participants
  hours
    number analyzed (Participants) | 21
    (all) | 14.7 (3.12)
Unaided Right PTA [Mean (Standard Deviation); unit: dB] — Pure Tone Average (PTA) assesses the average of hearing threshold levels at a set of specified frequencies. It is measured in decibels. Normal hearing is about 0-25 decibels for sounds in the normal speech frequency range. Population: Data is missing for one participant.
  dB
    PTA (avg 500, 1000, 2000): number analyzed (Participants) | 24
    PTA (avg 500, 1000, 2000) | 94.0 (23.8)
    High Frequency PTA: number analyzed (Participants) | 24
    High Frequency PTA | 98.8 (23.2)
    Low Frequency PTA: number analyzed (Participants) | 24
    Low Frequency PTA | 80.5 (28.3)
Unaided Left PTA [Mean (Standard Deviation); unit: dB] — Pure Tone Average (PTA) assesses the average of hearing threshold levels at a set of specified frequencies. It is measured in decibels. Normal hearing is about 0-25 decibels for sounds in the normal speech frequency range. Population: Data is missing for one participant (could not be collected)
  dB
    PTA (avg 500, 1000, 2000): number analyzed (Participants) | 24
    PTA (avg 500, 1000, 2000) | 94.0 (24.1)
    High Frequency PTA: number analyzed (Participants) | 24
    High Frequency PTA | 99.3 (23.5)
    Low Frequency PTA: number analyzed (Participants) | 24
    Low Frequency PTA | 77.0 (33.5)
PTA: Cochlear Implant Alone [Mean (Standard Deviation); unit: dB] — Pure Tone Average (PTA) assesses the average of hearing threshold levels at a set of specified frequencies. It is measured in decibels. Normal hearing is about 0-25 decibels for sounds in the normal speech frequency range. Population: Data could not be collected for 3 participants.
  dB
    PTA (avg 500, 1000, 2000): number analyzed (Participants) | 22
    PTA (avg 500, 1000, 2000) | 29.5 (5.67)
    High Frequency PTA: number analyzed (Participants) | 22
    High Frequency PTA | 28.2 (4.87)
    Low Frequency PTA: number analyzed (Participants) | 22
    Low Frequency PTA | 31.1 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Cochlear Implant: Signal to Noise Ratio (SNR) Threshold Obtained From IEEE (Speech Perception in Noise Test) Sentence in Noise Test.
Description: The IEEE test allows a researcher to evaluate how well a subject understands sentences in noisy situations. Primary Outcome #1 will assess how well the listener can hear with his/her cochlear implant. The listener will be tested without a contralateral device versus also wearing a contralateral device while listening to sentences coming from various directions along with competing noise coming from various directions. The directions of the sentences or noise are as follows:
  * Omni: from all directions
  * Ipsi: the same side
  * Front
  * Contra: Contralateral, from the opposite side of the implant Visits are flexible, based on participant preference and may be completed any time between enrollment and end of study. Testing takes about 12 minutes.
Time Frame: 12 minutes
Population: One participant did not have data collected while wearing the contralateral device. Data is only available for 5 participants in the "No Contralateral Device" group. The PI has left the institution and multiple attempts to contact the PI or ascertain why only 5 participants were assessed for this group have been unsuccessful. This is the only data that can be provided.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- No Contralateral Device (Cochlear Implant Alone): Subject only uses the cochlear implant; hearing on the contralateral side is unaided.
  Cochlear Implant Alone: No hearing device on contralateral ear
- Cochlear Implant and Contralateral Device: Subject wears a contralateral device
Arm/Group | No Contralateral Device (Cochlear Implant Alone) | Cochlear Implant and Contralateral Device
Number analyzed (Participants) | 5 | 19
ratio
  CI, Ipsi Speech, Omni Noise | 8.45 (11.4) | 10.4 (9.5)
  CI, Contra Speech, Ipsi Noise | 21.2 (6.99) | 22.2 (6.17)
  CI, Contra Speech, Omni Noise | 15.5 (8.85) | 15.9 (7.73)
  CI, Front Speech, Front Noise | 15.8 (7.04) | 17.1 (6.94)
  CI, Front Speech, Omni Noise | 8.85 (5.95) | 12.6 (8.27)

2. Primary Outcome: CI CROS: Signal to Noise Ratio (SNR) Threshold Obtained From IEEE (Speech Perception in Noise Test) Sentence in Noise Test.
Description: The IEEE test allows a researcher to evaluate how well a subject understands sentences in noisy situations. Primary Outcome #2 will assess how well the listener can hear wearing his/her cochlear implant and a CROS (Contralateral Routing of Signals device). A CROS is a device on the opposite ear that sends the nose to the cochlear implant. The listener will be tested without a contralateral device versus also wearing a contralateral device while listening to sentences coming from various directions along with competing noise coming from various directions. The directions of the sentences or noise are as follows:
  * Omni: from all directions
  * Ipsi: the same side
  * Front
  * Contra: Contralateral, from the opposite side of the implant Visits are flexible, based on participant preference and may be completed any time between enrollment and end of study. Testing takes about 12 minutes.
Time Frame: 12 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- No Contralateral Device (Cochlear Implant and CROS): Cochlear Implant and CROS Subject wears the CROS device on the contralateral side of the cochlear implant. Subject will use a clinic-loaned CROS device.
- Contralateral Device (Cochlear Implant and CROS): Cochlear Implant and CROS plus contralateral device.
Arm/Group | No Contralateral Device (Cochlear Implant and CROS) | Contralateral Device (Cochlear Implant and CROS)
Number analyzed (Participants) | 5 | 19
ratio
  CICROS, Ipsi Speech, Omni Noise | 9.7 (7.17) | 13.7 (8.92)
  CICROS, Contra Speech, Ipsi Noise | 12.9 (10.3) | 16.6 (7.65)
  CICROS, Contra Speech, Omni | 9.9 (9.96) | 13.1 (8.2)
  CICROS, Front Speech, Front Noise | 15.3 (6.29) | 16.0 (7.26)
  CICROS, Front Speech, Omni Noise | 10.7 (4.65) | 13.5 (8.5)

3. Primary Outcome: CI HA: Signal to Noise Ratio (SNR) Threshold Obtained From IEEE (Speech Perception in Noise Test) Sentence in Noise Test.
Description: The IEEE test allows a researcher to evaluate how well a subject understands sentences in noisy situations. Primary Outcome #3 will assess how well the listener can hear wearing his/her cochlear implant and hearing aid. The listener will be tested without a contralateral device versus also wearing a contralateral device while listening to sentences coming from various directions along with competing noise coming from various directions. The directions of the sentences or noise are as follows:
  * Omni: from all directions
  * Ipsi: the same side
  * Front
  * Contra: Contralateral, from the opposite side of the implant Visits are flexible, based on participant preference and may be completed any time between enrollment and end of study. Testing takes about 12 minutes.
Time Frame: 12 minutes
Population: Data could not be collected for one participant while wearing the Contralateral Device for condition "CIHA, Contra Speech, Omni Noise". Data is only available for 5 participants in the "No Contralateral Device" group. The PI has left the institution and multiple attempts to contact the PI or ascertain why only 5 participants were assessed for this group have been unsuccessful. This is the only data that can be provided.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- No Contralateral Device (Cochlear Implant and Hearing Aid): Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests.
  Hearing Aid: Advanced Bionics Naida hearing aid
- Contralateral Device (Cochlear Implant and Hearing Aid): Subject wears a hearing aid on the contralateral side of the cochlear implant. Subject will use a clinic-loaned Naida hearing aid for listening tests.
  Subject wears a Contralateral Device
Arm/Group | No Contralateral Device (Cochlear Implant and Hearing Aid) | Contralateral Device (Cochlear Implant and Hearing Aid)
Number analyzed (Participants) | 5 | 20
ratio
  CIHA, Ipsi Speech, Omni Noise | 8.62 (10.5) | 9.05 (7.06)
  CIHA, Contra Speech, Ipsi Noise | 16.4 (8.19) | 16.9 (8.44)
  CIHA, Contra Speech, Omni Noise: number analyzed (Participants) | 5 | 19
  CIHA, Contra Speech, Omni Noise | 11.6 (10.1) | 11.5 (8.17)
  CIHA, Front Speech, Front Noise | 14.0 (6.78) | 14.6 (6.62)
  CIHA, Front Speech, Omni Noise | 8.65 (6.67) | 9.51 (7.49)

ADVERSE EVENTS:
Time Frame: 5 Days
Description: However, if a subject experiences an adverse event requiring medical attention, the patient will be offered treatment at the Otolaryngology Outpatient Clinic.
  Any adverse events and/or Unanticipated Adverse Events will be treated using the standard of care for the specific problem.
Arm/Group | Cochlear Implant and Hearing Aid | Cochlear Implant Alone | Cochlear Implant and CROS
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
A questionnaire related to listening effort and acceptability ratings was removed from the study and not collected. Outcome measures related to this questionnaire were not collected and have been removed from the record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03867396/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT03867396/ICF_001.pdf